CLINICAL TRIAL: NCT00800163
Title: Emergency Department Physician Activation of the Catheterization Laboratory and Immediate Transfer to an Immediately Available Catheterization Lab Reduce Door-to-Balloon Time in ST-Elevation Myocardial Infarction
Brief Title: Improving Door-to-Balloon Time in STEMI
Acronym: EHART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Francis Hospitals & Health Centers (Other)
Responsible Party: Umesh N. Khot, M.D., Indiana Heart Physicians/St. Francis Heart Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: St. Francis Heart Center-EHART
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2008-11

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ED Physician Activation/Immediate Transfer (Experimental)
  Interventions: Other: ED Activation/Immediate Transfer

INTERVENTIONS:
Other: ED Activation/Immediate Transfer — ED Physician Activation and Immediate Transfer Protocol - see Circulation. 2007;116:67-76

SUMMARY:
The investigators prospectively determined the impact on median door-to-balloon time of a protocol mandating (1) emergency department physician activation of the catheterization lab and (2) immediate transfer of the patient to an immediately available catheterization lab by an in-house transfer team consisting of an emergency department nurse, a critical care unit nurse, and a chest pain unit nurse.

DETAILED DESCRIPTION:
Please see Circulation. 2007;116:67-76

ELIGIBILITY:
Primary Study Inclusion Criteria:

* ST-elevation myocardial infarction patients who undergo percutaneous intervention within 24 hours of ED arrival

Exclusion Criteria:

* Patients who are inpatients

A registry of all patients who undergo emergency cardiac catheterization irrespective of etiology is maintained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2005-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Door-to-Balloon Time | 24 hours

SECONDARY OUTCOMES:
Infarct Size | 48 hours
In-Hospital Mortality | ~ 7 days (during index hospitalization)
Hospital Length of Stay | ~2-7 days (during index hospitalization)
Hospital Costs | ~2-7 days (during Index Hospitalization) and One Year Followup

CONTACTS AND LOCATIONS:
Overall Officials: Umesh N Khot, M.D., Principal Investigator — Indiana Heart Physicians/St. Francis Heart Center
Locations (1):
- St. Francis Heart Center, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Khot UN, Johnson ML, Ramsey C, Khot MB, Todd R, Shaikh SR, Berg WJ. Emergency department physician activation of the catheterization laboratory and immediate transfer to an immediately available catheterization laboratory reduce door-to-balloon time in ST-elevation myocardial infarction. Circulation. 2007 Jul 3;116(1):67-76. doi: 10.1161/CIRCULATIONAHA.106.677401. Epub 2007 Jun 11. PMID 17562960
- [Derived] Khot UN, Johnson-Wood ML, Geddes JB, Ramsey C, Khot MB, Taillon H, Todd R, Shaikh SR, Berg WJ. Financial impact of reducing door-to-balloon time in ST-elevation myocardial infarction: a single hospital experience. BMC Cardiovasc Disord. 2009 Jul 26;9:32. doi: 10.1186/1471-2261-9-32. PMID 19631001